CLINICAL TRIAL: NCT06682663
Title: Evaluation of the Effect of Live Streaming Exercise on the Improvement of Hepatic Steatosis and Fibrosis in Pregnant Women with MASLD and Its Study Based on the Liver-gut Axis Mechanism.
Brief Title: Impact of Live Streaming Exercise on Liver Health in MASLD Pregnant Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Beijing Friendship Hospital (Other); W.F. Maternal and Child Health Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00001052-24122
Record Dates: First submitted 2024-11-06; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Dysfunction-associated Steatotic Liver Disease
Keywords: Randomized Controlled Trial; Live streaming exercise

STUDY DESIGN:
Intervention Model Description: The study will randomize eligible MASLD pregnant women into two groups: a control group and an intervention group. The control group will receive standard prenatal care, while the intervention group will receive supervised exercise guidance starting from the 14th week of pregnancy and continuing through the 36+6th week. Quality control, data collection, and biological sample collection will be conducted throughout the intervention period.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Live Streaming Exercise (Experimental): Live Streaming Exercise:Conduct supervised exercise guidance interventions from the 14th week of pregnancy and continuing through the 36+6th week.
  Interventions: Behavioral: Live Streaming Exercise
- Regular care (No Intervention): Regular care:health education.

INTERVENTIONS:
Behavioral: Live Streaming Exercise — Participants try to achieve 150 minutes of moderate-vigorous training per week. The exercise program includes live streaming exercise by trained health professionals, including pregnancy-specific exercises, with professional pregnancy trainers to provide guidance and support when needed.
  Arms: Live Streaming Exercise

SUMMARY:
Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD) is a clinical and pathological syndrome characterized primarily by excessive intracellular fat accumulation in the liver, excluding alcohol-related and other specific causes. Recent research has identified an association between MASLD and an increased risk of pregnancy-related complications and adverse pregnancy outcomes, including gestational diabetes, preeclampsia, preterm birth, and large-for-gestational-age infants. MASLD in pregnant women poses multiple risks to maternal and infant health. Regular physical exercise during pregnancy has been shown to effectively reduce the incidence of pregnancy complications and adverse outcomes, while also alleviating hepatic steatosis and fibrosis. This study is a randomized controlled trial aimed at exploring the feasibility and effectiveness of online exercise interventions for pregnant women with MASLD, as well as conducting a cost-effectiveness analysis and investigating the underlying physiological mechanisms based on the liver-gut axis. The findings are intended to provide scientific evidence and practical recommendations for managing pregnancy health and intervening in MASLD during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy;
2. Gestational age ≤10-13+6 weeks at enrollment;
3. Age between 20 and 45 years;
4. Patients diagnosed with MASLD;
5. Signed informed consent.

Exclusion Criteria:

1. Cervical length ≤ 25 mm;
2. History of threatened abortion;
3. Exercise contraindications or doctor advice not to exercise during pregnancy;
4. Current or previous use of drugs that affect body weight (such as hormones);
5. Patients with chronic hepatitis virus or other chronic liver diseases, excluding MASLD;
6. Non-natural conception or infertility treatment;
7. Any previous medication for hypertension, diabetes, heart disease, kidney disease, systemic lupus erythematosus, thyroid disease or mental illness;
8. Participating in other pregnancy intervention research projects.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Liver steatosis | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  LiSA, by Hepatus, Mindray, China；
Liver stiffness measurement | Changes from the 14th week to 36 weeks +6 days of pregnancy
  E, by Hepatus, Mindray, China

SECONDARY OUTCOMES:
Gestational weight change | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  weight changes in kilograms
Incidence of pregnancy-related complications including gestational diabetes mellitus, gestational hypertension and related diseases | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  All diagnoses according to the guidelines.
Changes in fasting serum lipids(TG, TC, LDL, HDL) | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  All data with the routine health check-up.
Changes in fasting blood glucose | Changes from the 14th week to 36 weeks +6 days of pregnancy
  with the routine check-up
Changes in blood pressure | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  Both systolic and diastolic blood pressure are measured
Changes in alanine aminotransferase (ALT) | Changes from the 14th week to 36 weeks +6 days of pregnancy
Changes in aspartate aminotransferase (AST) | Changes from the 14th week to 36 weeks + 6 days of pregnancy
Maternal physical activity | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  physical activity, which collected by International Physical Activity Questionnaire Short Form，IPAQ-SF
Maternal sleep quality | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  sleep quality, which collected by Pittsburgh Sleep Quality Questionnaire
Maternal mental health | Changes from the 14th week to 36 weeks + 6 days of pregnancy
  mental health, which collected by Generalized Anxiety Disorder-7 questionnaire， Edinburgh Pregnancy Depression Scale and Patient Health Questionnaire-9 items
Fetal height and weight | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  fetal height and weight, measured by ultrasonic, height in cm and weight in kg
Height and weight at birth | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  height, weight at birth,height measured with a rangefinder and weight measured with a scale,height in cm and weight in kg
Baby's Apgar Score | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  Apgar score，measured by clinical diagnosis
Preterm birth | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  preterm birth,clinical diagnosis
Small gestational week | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  small gestational week,clinical diagnosis
Large gestational week | fetal data were collected from gestational week 14 to 36 week +6 days, other data collected on the delivery.
  large gestational week,clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Hui Wang, Ph.D, Principal Investigator — Peking University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630
- [Background] Zhou F, Zhou J, Wang W, Zhang XJ, Ji YX, Zhang P, She ZG, Zhu L, Cai J, Li H. Unexpected Rapid Increase in the Burden of NAFLD in China From 2008 to 2018: A Systematic Review and Meta-Analysis. Hepatology. 2019 Oct;70(4):1119-1133. doi: 10.1002/hep.30702. PMID 31070259
- [Background] Younossi ZM, Koenig AB, Abdelatif D, Fazel Y, Henry L, Wymer M. Global epidemiology of nonalcoholic fatty liver disease-Meta-analytic assessment of prevalence, incidence, and outcomes. Hepatology. 2016 Jul;64(1):73-84. doi: 10.1002/hep.28431. Epub 2016 Feb 22. PMID 26707365
- [Background] Qian Y, Zhang Y, Fan X, Yan H, Li X, Fan Y, Song Y, Ma S, Hu Z, Gao X, Yang J. Nonalcoholic Fatty Liver Disease and Adverse Pregnancy Outcomes in Women With Normal Prepregnant Weight. J Clin Endocrinol Metab. 2023 Jan 17;108(2):463-471. doi: 10.1210/clinem/dgac567. PMID 36181486
- [Background] Lee SM, Cho GJ, Wi WY, Norwitz ER, Koo BK, Lee J, Jung YM, Kwak SH, Park CW, Jun JK, Joo SK, Oh MJ, Kim W, Park JS. Metabolic dysfunction-associated fatty liver disease as a risk factor for adverse outcomes in subsequent pregnancy: a nationwide cohort study. Hepatol Int. 2023 Apr;17(2):367-376. doi: 10.1007/s12072-022-10458-w. Epub 2022 Dec 21. PMID 36542262
- [Background] Chai TY, Byth K, George J, Pasupathy D, Cheung NW. Elevated Hepatic Steatosis Index is Associated with the Development of Adverse Maternal, but Not Adverse Neonatal, Outcomes: A Retrospective Cohort Study. Int J Womens Health. 2023 Apr 13;15:589-598. doi: 10.2147/IJWH.S399085. eCollection 2023. PMID 37077282
- [Background] El Jamaly H, Eslick GD, Weltman M. Systematic review with meta-analysis: Non-alcoholic fatty liver disease and the association with pregnancy outcomes. Clin Mol Hepatol. 2022 Jan;28(1):52-66. doi: 10.3350/cmh.2021.0205. Epub 2021 Sep 17. PMID 34530527
- [Background] Sarkar M, Grab J, Dodge JL, Gunderson EP, Rubin J, Irani RA, Cedars M, Terrault N. Non-alcoholic fatty liver disease in pregnancy is associated with adverse maternal and perinatal outcomes. J Hepatol. 2020 Sep;73(3):516-522. doi: 10.1016/j.jhep.2020.03.049. Epub 2020 Jun 9. PMID 32531415
- [Background] Jung YM, Lee SM, Hong S, Koo JN, Oh IH, Kim BJ, Kim SM, Kim SY, Kim GM, Kyung Joo S, Shin S, Norwitz ER, Park CW, Jun JK, Kim W, Park JS. The risk of pregnancy-associated hypertension in women with nonalcoholic fatty liver disease. Liver Int. 2020 Oct;40(10):2417-2426. doi: 10.1111/liv.14563. Epub 2020 Jun 30. PMID 32558189
- [Background] Lee SM, Kwak SH, Koo JN, Oh IH, Kwon JE, Kim BJ, Kim SM, Kim SY, Kim GM, Joo SK, Koo BK, Shin S, Vixay C, Norwitz ER, Park CW, Jun JK, Kim W, Park JS. Non-alcoholic fatty liver disease in the first trimester and subsequent development of gestational diabetes mellitus. Diabetologia. 2019 Feb;62(2):238-248. doi: 10.1007/s00125-018-4779-8. Epub 2018 Nov 23. PMID 30470912
- [Background] Lee SM, Kim BJ, Koo JN, Norwitz ER, Oh IH, Kim SM, Kim SY, Kim GM, Kwak SH, Kim W, Joo SK, Shin S, Vixa C, Park CW, Jun JK, Park JS. Nonalcoholic fatty liver disease is a risk factor for large-for-gestational-age birthweight. PLoS One. 2019 Aug 26;14(8):e0221400. doi: 10.1371/journal.pone.0221400. eCollection 2019. PMID 31449538
- [Background] Herath RP, Siriwardana SR, Ekanayake CD, Abeysekara V, Kodithuwakku SUA, Herath HP. Non-alcoholic fatty liver disease and pregnancy complications among Sri Lankan women: A cross sectional analytical study. PLoS One. 2019 Apr 12;14(4):e0215326. doi: 10.1371/journal.pone.0215326. eCollection 2019. PMID 30978266
- [Background] Mousa N, Abdel-Razik A, Shams M, Sheta T, Zakaria S, Shabana W, Effat N, El-Diasty M, Abed S, Abd Elsalam M, Awad M, Salah M, El-Wakeel N, Deiab AG, Eldars W. Impact of non-alcoholic fatty liver disease on pregnancy. Br J Biomed Sci. 2018 Oct;75(4):197-199. doi: 10.1080/09674845.2018.1492205. Epub 2018 Aug 6. No abstract available. PMID 29943682
- [Background] Hagstrom H, Hoijer J, Ludvigsson JF, Bottai M, Ekbom A, Hultcrantz R, Stephansson O, Stokkeland K. Adverse outcomes of pregnancy in women with non-alcoholic fatty liver disease. Liver Int. 2016 Feb;36(2):268-74. doi: 10.1111/liv.12902. Epub 2015 Sep 9. PMID 26114995
- [Background] Cheng R, Wang L, Le S, Yang Y, Zhao C, Zhang X, Yang X, Xu T, Xu L, Wiklund P, Ge J, Lu D, Zhang C, Chen L, Cheng S. A randomized controlled trial for response of microbiome network to exercise and diet intervention in patients with nonalcoholic fatty liver disease. Nat Commun. 2022 May 10;13(1):2555. doi: 10.1038/s41467-022-29968-0. PMID 35538056
- [Background] Babu AF, Csader S, Lok J, Gomez-Gallego C, Hanhineva K, El-Nezami H, Schwab U. Positive Effects of Exercise Intervention without Weight Loss and Dietary Changes in NAFLD-Related Clinical Parameters: A Systematic Review and Meta-Analysis. Nutrients. 2021 Sep 8;13(9):3135. doi: 10.3390/nu13093135. PMID 34579012
- [Background] Romero-Gomez M, Zelber-Sagi S, Trenell M. Treatment of NAFLD with diet, physical activity and exercise. J Hepatol. 2017 Oct;67(4):829-846. doi: 10.1016/j.jhep.2017.05.016. Epub 2017 May 23. PMID 28545937
- [Background] Orci LA, Gariani K, Oldani G, Delaune V, Morel P, Toso C. Exercise-based Interventions for Nonalcoholic Fatty Liver Disease: A Meta-analysis and Meta-regression. Clin Gastroenterol Hepatol. 2016 Oct;14(10):1398-411. doi: 10.1016/j.cgh.2016.04.036. Epub 2016 May 4. PMID 27155553
- [Background] Oh S, Tsujimoto T, Kim B, Uchida F, Suzuki H, Iizumi S, Isobe T, Sakae T, Tanaka K, Shoda J. Weight-loss-independent benefits of exercise on liver steatosis and stiffness in Japanese men with NAFLD. JHEP Rep. 2021 Feb 10;3(3):100253. doi: 10.1016/j.jhepr.2021.100253. eCollection 2021 Jun. PMID 33898958
- [Background] Hashida R, Kawaguchi T, Bekki M, Omoto M, Matsuse H, Nago T, Takano Y, Ueno T, Koga H, George J, Shiba N, Torimura T. Aerobic vs. resistance exercise in non-alcoholic fatty liver disease: A systematic review. J Hepatol. 2017 Jan;66(1):142-152. doi: 10.1016/j.jhep.2016.08.023. Epub 2016 Sep 14. PMID 27639843
- [Background] Smart NA, King N, McFarlane JR, Graham PL, Dieberg G. Effect of exercise training on liver function in adults who are overweight or exhibit fatty liver disease: a systematic review and meta-analysis. Br J Sports Med. 2018 Jul;52(13):834-843. doi: 10.1136/bjsports-2016-096197. Epub 2016 Jun 17. PMID 27317790
- [Background] Zeng Y, Zhang X, Luo W, Sheng Y. Effect of exercise intervention on clinical parameters in patients with non-alcoholic fatty liver disease and type 2 diabetes mellitus: a meta-analysis of randomized controlled trials. Eur J Gastroenterol Hepatol. 2024 Jan 1;36(1):1-12. doi: 10.1097/MEG.0000000000002662. PMID 37942754
- [Background] Liu Y, Xie W, Li J, Ossowski Z. Effects of aerobic exercise on metabolic indicators and physical performance in adult NAFLD patients: A systematic review and network meta-analysis. Medicine (Baltimore). 2023 Apr 7;102(14):e33147. doi: 10.1097/MD.0000000000033147. PMID 37026928
- [Background] Nam H, Yoo JJ, Cho Y, Kang SH, Ahn SB, Lee HW, Jun DW, Song DS, Choi M. Effect of exercise-based interventions in nonalcoholic fatty liver disease: A systematic review with meta-analysis. Dig Liver Dis. 2023 Sep;55(9):1178-1186. doi: 10.1016/j.dld.2022.12.013. Epub 2023 Jan 16. PMID 36653265
- [Background] Clifton RG, Evans M, Cahill AG, Franks PW, Gallagher D, Phelan S, Pomeroy J, Redman LM, Van Horn L; LIFE-Moms Research Group. Design of lifestyle intervention trials to prevent excessive gestational weight gain in women with overweight or obesity. Obesity (Silver Spring). 2016 Feb;24(2):305-13. doi: 10.1002/oby.21330. Epub 2015 Dec 26. PMID 26708836
- [Background] Poston L, Bell R, Croker H, Flynn AC, Godfrey KM, Goff L, Hayes L, Khazaezadeh N, Nelson SM, Oteng-Ntim E, Pasupathy D, Patel N, Robson SC, Sandall J, Sanders TA, Sattar N, Seed PT, Wardle J, Whitworth MK, Briley AL; UPBEAT Trial Consortium. Effect of a behavioural intervention in obese pregnant women (the UPBEAT study): a multicentre, randomised controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):767-77. doi: 10.1016/S2213-8587(15)00227-2. Epub 2015 Jul 9. PMID 26165396
- [Background] Effect of diet and physical activity based interventions in pregnancy on gestational weight gain and pregnancy outcomes: meta-analysis of individual participant data from randomised trials. BMJ. 2017 Aug 23;358:j3991. doi: 10.1136/bmj.j3991. No abstract available. PMID 28835414
- [Background] Facchinetti F, Vijai V, Petrella E, Gambigliani Zoccoli S, Pignatti L, Di Cerbo L, Neri I. Food glycemic index changes in overweight/obese pregnant women enrolled in a lifestyle program: a randomized controlled trial. Am J Obstet Gynecol MFM. 2019 Aug;1(3):100030. doi: 10.1016/j.ajogmf.2019.100030. Epub 2019 Aug 5. PMID 33345794
- [Background] Bruno R, Petrella E, Bertarini V, Pedrielli G, Neri I, Facchinetti F. Adherence to a lifestyle programme in overweight/obese pregnant women and effect on gestational diabetes mellitus: a randomized controlled trial. Matern Child Nutr. 2017 Jul;13(3):e12333. doi: 10.1111/mcn.12333. Epub 2016 Sep 19. PMID 27647837
- [Background] Altazan AD, Redman LM, Burton JH, Beyl RA, Cain LE, Sutton EF, Martin CK. Mood and quality of life changes in pregnancy and postpartum and the effect of a behavioral intervention targeting excess gestational weight gain in women with overweight and obesity: a parallel-arm randomized controlled pilot trial. BMC Pregnancy Childbirth. 2019 Jan 29;19(1):50. doi: 10.1186/s12884-019-2196-8. PMID 30696408
- [Background] Gascoigne EL, Webster CM, Honart AW, Wang P, Smith-Ryan A, Manuck TA. Physical activity and pregnancy outcomes: an expert review. Am J Obstet Gynecol MFM. 2023 Jan;5(1):100758. doi: 10.1016/j.ajogmf.2022.100758. Epub 2022 Sep 26. PMID 36174931
- [Background] Sanabria-Martinez G, Garcia-Hermoso A, Poyatos-Leon R, Gonzalez-Garcia A, Sanchez-Lopez M, Martinez-Vizcaino V. Effects of Exercise-Based Interventions on Neonatal Outcomes: A Meta-Analysis of Randomized Controlled Trials. Am J Health Promot. 2016 Mar;30(4):214-23. doi: 10.1177/0890117116639569. PMID 27404056
- [Background] Di Mascio D, Magro-Malosso ER, Saccone G, Marhefka GD, Berghella V. Exercise during pregnancy in normal-weight women and risk of preterm birth: a systematic review and meta-analysis of randomized controlled trials. Am J Obstet Gynecol. 2016 Nov;215(5):561-571. doi: 10.1016/j.ajog.2016.06.014. Epub 2016 Jun 16. PMID 27319364
- [Background] Physical Activity and Exercise During Pregnancy and the Postpartum Period: ACOG Committee Opinion, Number 804. Obstet Gynecol. 2020 Apr;135(4):e178-e188. doi: 10.1097/AOG.0000000000003772. PMID 32217980
- [Background] Mottola MF, Davenport MH, Ruchat SM, Davies GA, Poitras VJ, Gray CE, Jaramillo Garcia A, Barrowman N, Adamo KB, Duggan M, Barakat R, Chilibeck P, Fleming K, Forte M, Korolnek J, Nagpal T, Slater LG, Stirling D, Zehr L. 2019 Canadian guideline for physical activity throughout pregnancy. Br J Sports Med. 2018 Nov;52(21):1339-1346. doi: 10.1136/bjsports-2018-100056. PMID 30337460
- [Background] Evenson KR, Barakat R, Brown WJ, Dargent-Molina P, Haruna M, Mikkelsen EM, Mottola MF, Owe KM, Rousham EK, Yeo S. Guidelines for Physical Activity during Pregnancy: Comparisons From Around the World. Am J Lifestyle Med. 2014 Mar;8(2):102-121. doi: 10.1177/1559827613498204. PMID 25346651
- [Background] Simmons D, Jelsma JG, Galjaard S, Devlieger R, van Assche A, Jans G, Corcoy R, Adelantado JM, Dunne F, Desoye G, Harreiter J, Kautzky-Willer A, Damm P, Mathiesen ER, Jensen DM, Andersen LL, Lapolla A, Dalfra M, Bertolotto A, Wender-Ozegowska E, Zawiejska A, Hill D, Rebollo P, Snoek FJ, van Poppel MN. Results From a European Multicenter Randomized Trial of Physical Activity and/or Healthy Eating to Reduce the Risk of Gestational Diabetes Mellitus: The DALI Lifestyle Pilot. Diabetes Care. 2015 Sep;38(9):1650-6. doi: 10.2337/dc15-0360. Epub 2015 Jun 25. PMID 26112044
- [Background] Dodd JM, Deussen AR, Louise J. Optimising gestational weight gain and improving maternal and infant health outcomes through antenatal dietary, lifestyle and physical activity advice: the OPTIMISE randomised controlled trial protocol. BMJ Open. 2018 Feb 20;8(2):e019583. doi: 10.1136/bmjopen-2017-019583. PMID 29463591
- [Background] Pauley AM, Hohman E, Savage JS, Rivera DE, Guo P, Leonard KS, Symons Downs D. Gestational Weight Gain Intervention Impacts Determinants of Healthy Eating and Exercise in Overweight/Obese Pregnant Women. J Obes. 2018 Oct 1;2018:6469170. doi: 10.1155/2018/6469170. eCollection 2018. PMID 30364005
- [Background] Vinter CA, Tanvig MH, Christensen MH, Ovesen PG, Jorgensen JS, Andersen MS, McIntyre HD, Jensen DM. Lifestyle Intervention in Danish Obese Pregnant Women With Early Gestational Diabetes Mellitus According to WHO 2013 Criteria Does Not Change Pregnancy Outcomes: Results From the LiP (Lifestyle in Pregnancy) Study. Diabetes Care. 2018 Oct;41(10):2079-2085. doi: 10.2337/dc18-0808. Epub 2018 Jul 30. PMID 30061318
- [Background] McGiveron A, Foster S, Pearce J, Taylor MA, McMullen S, Langley-Evans SC. Limiting antenatal weight gain improves maternal health outcomes in severely obese pregnant women: findings of a pragmatic evaluation of a midwife-led intervention. J Hum Nutr Diet. 2015 Jan;28 Suppl 1:29-37. doi: 10.1111/jhn.12240. Epub 2014 May 9. PMID 24809211
- [Background] Liu J, Wilcox S, Hutto B, Turner-McGrievy G, Wingard E. Effects of a lifestyle intervention on postpartum weight retention among women with elevated weight. Obesity (Silver Spring). 2022 Jul;30(7):1370-1379. doi: 10.1002/oby.23449. Epub 2022 Jun 20. PMID 35722816
- [Background] Dodd JM, Cramp C, Sui Z, Yelland LN, Deussen AR, Grivell RM, Moran LJ, Crowther CA, Turnbull D, McPhee AJ, Wittert G, Owens JA, Robinson JS; LIMIT Randomised Trial Group. The effects of antenatal dietary and lifestyle advice for women who are overweight or obese on maternal diet and physical activity: the LIMIT randomised trial. BMC Med. 2014 Oct 13;12:161. doi: 10.1186/s12916-014-0161-y. PMID 25315237
- [Background] Wilcox S, Liu J, Turner-McGrievy GM, Boutte AK, Wingard E. Effects of a behavioral intervention on physical activity, diet, and health-related quality of life in pregnant women with elevated weight: results of the HIPP randomized controlled trial. Int J Behav Nutr Phys Act. 2022 Dec 9;19(1):145. doi: 10.1186/s12966-022-01387-w. PMID 36494702
- [Background] Bisson M, Almeras N, Dufresne SS, Robitaille J, Rheaume C, Bujold E, Frenette J, Tremblay A, Marc I. A 12-Week Exercise Program for Pregnant Women with Obesity to Improve Physical Activity Levels: An Open Randomised Preliminary Study. PLoS One. 2015 Sep 16;10(9):e0137742. doi: 10.1371/journal.pone.0137742. eCollection 2015. PMID 26375471
- [Background] Wang C, Wei Y, Zhang X, Zhang Y, Xu Q, Sun Y, Su S, Zhang L, Liu C, Feng Y, Shou C, Guelfi KJ, Newnham JP, Yang H. A randomized clinical trial of exercise during pregnancy to prevent gestational diabetes mellitus and improve pregnancy outcome in overweight and obese pregnant women. Am J Obstet Gynecol. 2017 Apr;216(4):340-351. doi: 10.1016/j.ajog.2017.01.037. Epub 2017 Feb 1. PMID 28161306
- [Background] Li HT, Xue M, Hellerstein S, Cai Y, Gao Y, Zhang Y, Qiao J, Blustein J, Liu JM. Association of China's universal two child policy with changes in births and birth related health factors: national, descriptive comparative study. BMJ. 2019 Aug 21;366:l4680. doi: 10.1136/bmj.l4680. PMID 31434652
- [Background] Ferrara A, Hedderson MM, Brown SD, Ehrlich SF, Tsai AL, Feng J, Galarce M, Marcovina S, Catalano P, Quesenberry CP. A telehealth lifestyle intervention to reduce excess gestational weight gain in pregnant women with overweight or obesity (GLOW): a randomised, parallel-group, controlled trial. Lancet Diabetes Endocrinol. 2020 Jun;8(6):490-500. doi: 10.1016/S2213-8587(20)30107-8. PMID 32445736
- [Background] Deruelle P, Lelorain S, Deghilage S, Couturier E, Guilbert E, Berveiller P, Senat MV, Vayssiere C, Sentilhes L, Perrotin F, Gallot D, Chauleur C, Sananes N, Roth E, Luton D, Caputo M, Lorio E, Chatelet C, Couster J, Timbely O, Doret-Dion M, Duhamel A, Pigeyre M. Rationale and design of ePPOP-ID: a multicenter randomized controlled trial using an electronic-personalized program for obesity in pregnancy to improve delivery. BMC Pregnancy Childbirth. 2020 Oct 7;20(1):602. doi: 10.1186/s12884-020-03288-x. PMID 33028261
- [Background] Hayman M, Reaburn P, Browne M, Vandelanotte C, Alley S, Short CE. Feasibility, acceptability and efficacy of a web-based computer-tailored physical activity intervention for pregnant women - the Fit4Two randomised controlled trial. BMC Pregnancy Childbirth. 2017 Mar 23;17(1):96. doi: 10.1186/s12884-017-1277-9. PMID 28335767
- [Background] Yu H, Santos-Rocha R, Radziminski L, Jastrzebski Z, Bonislawska I, Szwarc A, Szumilewicz A. Effects of 8-Week Online, Supervised High-Intensity Interval Training on the Parameters Related to the Anaerobic Threshold, Body Weight, and Body Composition during Pregnancy: A Randomized Controlled Trial. Nutrients. 2022 Dec 11;14(24):5279. doi: 10.3390/nu14245279. PMID 36558438
- [Background] Mazzotti A, Caletti MT, Brodosi L, Di Domizio S, Forchielli ML, Petta S, Bugianesi E, Bianchi G, Marchesini G. An internet-based approach for lifestyle changes in patients with NAFLD: Two-year effects on weight loss and surrogate markers. J Hepatol. 2018 Nov;69(5):1155-1163. doi: 10.1016/j.jhep.2018.07.013. Epub 2018 Oct 2. PMID 30290973
- [Background] Petroni ML, Colosimo S, Brodosi L, Armandi A, Bertini F, Montesi D, Bugianesi E, Marchesini G. Long-term follow-up of web-based and group-based behavioural intervention in NAFLD in a real world clinical setting. Aliment Pharmacol Ther. 2024 Jan;59(2):249-259. doi: 10.1111/apt.17768. Epub 2023 Oct 16. PMID 37843741
- [Background] Kwon OY, Lee MK, Lee HW, Kim H, Lee JS, Jang Y. Mobile App-Based Lifestyle Coaching Intervention for Patients With Nonalcoholic Fatty Liver Disease: Randomized Controlled Trial. J Med Internet Res. 2024 Feb 15;26:e49839. doi: 10.2196/49839. PMID 38358794
- [Background] Dodd JM, Louise J, Cramp C, Grivell RM, Moran LJ, Deussen AR. Evaluation of a smartphone nutrition and physical activity application to provide lifestyle advice to pregnant women: The SNAPP randomised trial. Matern Child Nutr. 2018 Jan;14(1):e12502. doi: 10.1111/mcn.12502. Epub 2017 Aug 24. PMID 28836373
- [Background] Zheng Y, Wang W, Zhong Y, Wu F, Zhu Z, Tham YC, Lamoureux E, Xiao L, Zhu E, Liu H, Jin L, Liang L, Luo L, He M, Morgan I, Congdon N, Liu Y. A Peer-to-Peer Live-Streaming Intervention for Children During COVID-19 Homeschooling to Promote Physical Activity and Reduce Anxiety and Eye Strain: Cluster Randomized Controlled Trial. J Med Internet Res. 2021 Apr 30;23(4):e24316. doi: 10.2196/24316. PMID 33882021
- [Background] Tian R, Yin R, Gan F. Exploring public attitudes toward live-streaming fitness in China: A sentiment and content analysis of China's social media Weibo. Front Public Health. 2022 Nov 3;10:1027694. doi: 10.3389/fpubh.2022.1027694. eCollection 2022. PMID 36408048
- [Background] Rinella ME. Nonalcoholic fatty liver disease: a systematic review. JAMA. 2015 Jun 9;313(22):2263-73. doi: 10.1001/jama.2015.5370. PMID 26057287
- [Background] Houttu V, Boulund U, Grefhorst A, Soeters MR, Pinto-Sietsma SJ, Nieuwdorp M, Holleboom AG. The role of the gut microbiome and exercise in non-alcoholic fatty liver disease. Therap Adv Gastroenterol. 2020 Sep 15;13:1756284820941745. doi: 10.1177/1756284820941745. eCollection 2020. PMID 32973925
- [Background] Kim KH, Kim SH, Min YK, Yang HM, Lee JB, Lee MS. Acute exercise induces FGF21 expression in mice and in healthy humans. PLoS One. 2013 May 7;8(5):e63517. doi: 10.1371/journal.pone.0063517. Print 2013. PMID 23667629
- [Background] Dolegowska K, Marchelek-Mysliwiec M, Nowosiad-Magda M, Slawinski M, Dolegowska B. FGF19 subfamily members: FGF19 and FGF21. J Physiol Biochem. 2019 Jun;75(2):229-240. doi: 10.1007/s13105-019-00675-7. Epub 2019 Mar 29. PMID 30927227
- [Background] Tucker B, Li H, Long X, Rye KA, Ong KL. Fibroblast growth factor 21 in non-alcoholic fatty liver disease. Metabolism. 2019 Dec;101:153994. doi: 10.1016/j.metabol.2019.153994. Epub 2019 Oct 28. PMID 31672443
- [Background] Liu W, Sun C, Yan Y, Cao H, Niu Z, Shen S, Liu S, Wu Y, Li Y, Hui L, Li Y, Zhao L, Hu C, Ding Q, Jiang J, Ying H. Hepatic P38 Activation Modulates Systemic Metabolism Through Fgf21-Mediated Interorgan Communication. Diabetes. 2021 Oct 21:db210240. doi: 10.2337/db21-0240. Online ahead of print. PMID 34957482
- [Background] Zarei M, Pizarro-Delgado J, Barroso E, Palomer X, Vazquez-Carrera M. Targeting FGF21 for the Treatment of Nonalcoholic Steatohepatitis. Trends Pharmacol Sci. 2020 Mar;41(3):199-208. doi: 10.1016/j.tips.2019.12.005. Epub 2020 Jan 21. PMID 31980251
- [Background] Geng L, Liao B, Jin L, Huang Z, Triggle CR, Ding H, Zhang J, Huang Y, Lin Z, Xu A. Exercise Alleviates Obesity-Induced Metabolic Dysfunction via Enhancing FGF21 Sensitivity in Adipose Tissues. Cell Rep. 2019 Mar 5;26(10):2738-2752.e4. doi: 10.1016/j.celrep.2019.02.014. PMID 30840894
- [Background] Takahashi A, Abe K, Fujita M, Hayashi M, Okai K, Ohira H. Simple resistance exercise decreases cytokeratin 18 and fibroblast growth factor 21 levels in patients with nonalcoholic fatty liver disease: A retrospective clinical study. Medicine (Baltimore). 2020 May 29;99(22):e20399. doi: 10.1097/MD.0000000000020399. PMID 32481431
- [Background] Stine JG, Welles JE, Keating S, Hussaini Z, Soriano C, Heinle JW, Geyer N, Chinchilli VM, Loomba R, Kimball SR. Serum Fibroblast Growth Factor 21 Is Markedly Decreased following Exercise Training in Patients with Biopsy-Proven Nonalcoholic Steatohepatitis. Nutrients. 2023 Mar 20;15(6):1481. doi: 10.3390/nu15061481. PMID 36986211
- [Background] Gao Y, Zhang W, Zeng LQ, Bai H, Li J, Zhou J, Zhou GY, Fang CW, Wang F, Qin XJ. Exercise and dietary intervention ameliorate high-fat diet-induced NAFLD and liver aging by inducing lipophagy. Redox Biol. 2020 Sep;36:101635. doi: 10.1016/j.redox.2020.101635. Epub 2020 Jul 7. PMID 32863214
- [Background] Salminen A, Kauppinen A, Kaarniranta K. FGF21 activates AMPK signaling: impact on metabolic regulation and the aging process. J Mol Med (Berl). 2017 Feb;95(2):123-131. doi: 10.1007/s00109-016-1477-1. Epub 2016 Sep 27. PMID 27678528
- [Background] Mishra AK, Dubey V, Ghosh AR. Obesity: An overview of possible role(s) of gut hormones, lipid sensing and gut microbiota. Metabolism. 2016 Jan;65(1):48-65. doi: 10.1016/j.metabol.2015.10.008. Epub 2015 Nov 13. PMID 26683796
- [Background] Liu Y, Wang Y, Ni Y, Cheung CKY, Lam KSL, Wang Y, Xia Z, Ye D, Guo J, Tse MA, Panagiotou G, Xu A. Gut Microbiome Fermentation Determines the Efficacy of Exercise for Diabetes Prevention. Cell Metab. 2020 Jan 7;31(1):77-91.e5. doi: 10.1016/j.cmet.2019.11.001. Epub 2019 Nov 27. PMID 31786155
- [Background] Alisi A, Ceccarelli S, Panera N, Nobili V. Causative role of gut microbiota in non-alcoholic fatty liver disease pathogenesis. Front Cell Infect Microbiol. 2012 Oct 26;2:132. doi: 10.3389/fcimb.2012.00132. eCollection 2012. No abstract available. PMID 23112961
- [Background] Tremaroli V, Backhed F. Functional interactions between the gut microbiota and host metabolism. Nature. 2012 Sep 13;489(7415):242-9. doi: 10.1038/nature11552. PMID 22972297
- [Background] Nicoletti C. Age-associated changes of the intestinal epithelial barrier: local and systemic implications. Expert Rev Gastroenterol Hepatol. 2015;9(12):1467-9. doi: 10.1586/17474124.2015.1092872. Epub 2015 Sep 22. PMID 26395417
- [Background] Biagi E, Nylund L, Candela M, Ostan R, Bucci L, Pini E, Nikkila J, Monti D, Satokari R, Franceschi C, Brigidi P, De Vos W. Through ageing, and beyond: gut microbiota and inflammatory status in seniors and centenarians. PLoS One. 2010 May 17;5(5):e10667. doi: 10.1371/journal.pone.0010667. PMID 20498852
- [Background] Spencer MD, Hamp TJ, Reid RW, Fischer LM, Zeisel SH, Fodor AA. Association between composition of the human gastrointestinal microbiome and development of fatty liver with choline deficiency. Gastroenterology. 2011 Mar;140(3):976-86. doi: 10.1053/j.gastro.2010.11.049. Epub 2010 Dec 1. PMID 21129376
- [Background] Wang Z, Tang WH, Buffa JA, Fu X, Britt EB, Koeth RA, Levison BS, Fan Y, Wu Y, Hazen SL. Prognostic value of choline and betaine depends on intestinal microbiota-generated metabolite trimethylamine-N-oxide. Eur Heart J. 2014 Apr;35(14):904-10. doi: 10.1093/eurheartj/ehu002. Epub 2014 Feb 3. PMID 24497336
- [Background] Sayin SI, Wahlstrom A, Felin J, Jantti S, Marschall HU, Bamberg K, Angelin B, Hyotylainen T, Oresic M, Backhed F. Gut microbiota regulates bile acid metabolism by reducing the levels of tauro-beta-muricholic acid, a naturally occurring FXR antagonist. Cell Metab. 2013 Feb 5;17(2):225-35. doi: 10.1016/j.cmet.2013.01.003. PMID 23395169
- [Background] McMahan RH, Wang XX, Cheng LL, Krisko T, Smith M, El Kasmi K, Pruzanski M, Adorini L, Golden-Mason L, Levi M, Rosen HR. Bile acid receptor activation modulates hepatic monocyte activity and improves nonalcoholic fatty liver disease. J Biol Chem. 2013 Apr 26;288(17):11761-70. doi: 10.1074/jbc.M112.446575. Epub 2013 Mar 4. PMID 23460643
- [Background] Sinal CJ, Tohkin M, Miyata M, Ward JM, Lambert G, Gonzalez FJ. Targeted disruption of the nuclear receptor FXR/BAR impairs bile acid and lipid homeostasis. Cell. 2000 Sep 15;102(6):731-44. doi: 10.1016/s0092-8674(00)00062-3. PMID 11030617
- [Background] Swann JR, Want EJ, Geier FM, Spagou K, Wilson ID, Sidaway JE, Nicholson JK, Holmes E. Systemic gut microbial modulation of bile acid metabolism in host tissue compartments. Proc Natl Acad Sci U S A. 2011 Mar 15;108 Suppl 1(Suppl 1):4523-30. doi: 10.1073/pnas.1006734107. Epub 2010 Sep 13. PMID 20837534
- [Background] Leung C, Rivera L, Furness JB, Angus PW. The role of the gut microbiota in NAFLD. Nat Rev Gastroenterol Hepatol. 2016 Jul;13(7):412-25. doi: 10.1038/nrgastro.2016.85. Epub 2016 Jun 8. PMID 27273168
- [Background] Ye X, Sun P, Lao S, Wen M, Zheng R, Lin Y, Gan L, Fan X, Wang P, Li Z, Yan X, Zhao L. Fgf21-Dubosiella axis mediates the protective effects of exercise against NAFLD development. Life Sci. 2023 Dec 1;334:122231. doi: 10.1016/j.lfs.2023.122231. Epub 2023 Nov 5. PMID 37935276